CLINICAL TRIAL: NCT04193683
Title: The Effect Of Myofascial Release Technique On Respiratory Functions, Respiratory Muscle Strength and Endurance in Subjects With Short Hamstring Muscle
Brief Title: The Effect Of Myofascial Release Technique On Respiratory Parameters in Subjects With Short Hamstring Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: bvubcinar01
Record Dates: First submitted 2019-12-03; First posted 2019-12-10 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Hamstring Contractures
Keywords: Hamstring Muscle; Hamstring Shortness; Hamstring Stiffness; Myofascial Release Technique; Respiratory Functions; Respiratory Muscle Strength; Respiratory Muscle Endurance
MeSH Terms: interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham-Ultrasound (Sham Comparator): Intervention will include one session sham-ultrasound application to both lower extremities of participant. The total time will be 15 minutes.
  Interventions: Other: Sham-Ultrasound
- Myofascial Release Technique+Sham-Ultrasound (Experimental): In addition to one session sham-ultrasound, the intervention will include one session myofascial release technique to both lower extremities of participant. The total time will be 30 minutes.
  Interventions: Other: Myofascial Release Technique; Other: Sham-Ultrasound

INTERVENTIONS:
Other: Myofascial Release Technique — Myofascial release technique will bi applied bottom of the feet, back of the legs and hamstrings in both extremities. The practitioner will decide how long she should stay in a region according to the feeling of releasing in the tissue. The technique will be applied to a region at least 3 times.
  Arms: Myofascial Release Technique+Sham-Ultrasound
Other: Sham-Ultrasound — Sham-ultrasound will be applied to back of legs and thighs in both extremities without pressure and all parameters of the ultrasound device except the timer will be closed.

SUMMARY:
The aim of this study was to investigate the effect of myofascial release technique on rib cage mobility, respiratory function, respiratory muscle strength and endurance in patients with hamstring muscle shortness.

DETAILED DESCRIPTION:
Hamstring flexibility is important to maintain activities such as walking and running in daily life. Hamstring muscle shortness, commonly seen in the community, is a risk factor for many musculoskeletal pathologies. Clinical observations have shown that the shortness of the Hamstring muscle causes spinal malalignment. This deterioration of the spine alignment may adversely affect the rib cage expansion. Moreover, considering that the optimal length of the muscles provides optimal contraction, it was found that the spinal malalignment adversely affected the effective contraction of the diaphragm by changing the position of diaphragm. A different view is that, because the fascia functions as a single tissue surrounding the entire body, a restriction in the hamstring muscle can also cause a restriction in distal muscles such as diaphragm through the fascia.

There are many treatment methods used to increase the flexibility of the hamstring muscle. One of these methods is the myofascial release technique. In this technique, which targets both muscle and fascia, applying light and prolonged pressure provides the myo-fascial complex to reach its optimal length, resulting in the optimal function of the muscle. In our best knowledge, no study has evaluated the effect of myofascial release technique on respiratory parameters in patients with hamstring muscle shortness.

ELIGIBILITY:
Inclusion Criteria:

* more than 15 degrees knee flexion angle during popliteal angle test,
* no generalized joint laxity according to Beighton Criteria, and
* no musculoskeletal problems of lower extremities.

Exclusion Criteria:

* history of lower extremity and/or axial skeletal fracture;
* recent muscle, tendon injury in lower extremity;
* history of lumbal disc herniation, arthritic and/or inflammatory disease;
* obesity, diabetes and/or metabolic syndrome;
* history of surgery in the last month,
* using muscle relaxant medication in the last month;
* received manual therapy in the last month

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline Forced Vital Capacity (FVC) at 60 minutes | 60 minutes
  Respiratory Function Test
Change from baseline Forced Expiratory Volume in 1 second (FEV1) at 60 minutes | 60 minutes
  Respiratory Function Test
Change from baseline FEV1/FVC at 60 minutes | 60 minutes
  Respiratory Function Test
Change from baseline Peak Expiratory Flow (PEF) at 60 minutes | 60 minutes
  Respiratory Function Test
Change from baseline Forced expiratory flow over the middle one half of the FVC (FEF25-75%) at 60 minutes | 60 minutes
  Respiratory Function Test
Change from baseline maximum inspiratory pressure (MIP) at 60 minutes | 60 minutes
  Respiratory Muscle Strength Test
Change from baseline maximum expiratory pressure (MEP) at 60 minutes | 60 minutes
  Respiratory Muscle Strength Test
Change from baseline constant inspiratory threshold load test at 60 minutes | 60 minutes
  Respiratory Muscle Endurance Test

SECONDARY OUTCOMES:
Change from baseline axillary region chest circumference measurement during inspiration at 60 minutes | 60 minutes
  Chest Circumference Measurement
Change from baseline axillary region chest circumference measurement during expiration at 60 minutes | 60 minutes
  Chest Circumference Measurement
Change from baseline xiphoid region chest circumference measurement during inspiration at 60 minutes | 60 minutes
  Chest Circumference Measurement
Change from baseline xiphoid region chest circumference measurement during expiration at 60 minutes | 60 minutes
  Chest Circumference Measurement
Change from baseline subcostal region chest circumference measurement during inspiration at 60 minutes | 60 minutes
  Chest Circumference Measurement
Change from baseline subcostal region chest circumference measurement during expiration at 60 minutes | 60 minutes
  Chest Circumference Measurement
Change from baseline axillary region chest expansion test at 60 minutes | 60 minutes
  Chest Circumference Measurement
Change from baseline xiphoid region chest expansion test at 60 minutes | 60 minutes
  Chest Circumference Measurement
Change from baseline subcostal region chest expansion test at 60 minutes | 60 minutes
  Chest Circumference Measurement

CONTACTS AND LOCATIONS:
Overall Officials: Betül Çınar, Study Chair — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No